CLINICAL TRIAL: NCT06300996
Title: Spinal Cord Stimulation for the Treatment of Motor Deficits in People With Spinal Muscular Atrophy - Upper Limb Protocol
Brief Title: Spinal Cord Stimulation for the Treatment of Motor Deficits in People With Spinal Muscular Atrophy - Upper Limb
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Capogrosso (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor-Investigator, Marco Capogrosso, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY23110042
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Spinal Muscular Atrophy; Spinal Muscular Atrophy Type 3; Spinal Muscular Atrophy Type II; Spinal Muscular Atrophy 4; SMA
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Spinal muscular atrophy 4

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study performed to quantify variables that are predictive of the efficacy of spinal cord stimulation to improve motor control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): All patients will receive FDA-approved percutaneous spinal cord stimulation leads implanted in the cervical epidural (C4-T1 vertebra) space. The leads will be connected to external stimulators (either FDA-approved or human-grade research stimulator with safety features) during research activities.
  Interventions: Device: Spinal Cord Stimulator (Octopolar Medtronic Vectris Leads)

INTERVENTIONS:
Device: Spinal Cord Stimulator (Octopolar Medtronic Vectris Leads) — Spinal cord stimulation is FDA approved for treatment of pain. We are proposing utilizing the same technology to help restore motor control in people who have declining function due to the progression of SMA. These are 2-4 leads that are FDA-approved.

SUMMARY:
Spinal cord stimulation (SCS) has shown remarkable efficacy in restoring motor function in people with spinal cord injury by recruiting afferent input to enhance the responsiveness of spared neural circuits to residual cortical inputs. This pilot will test if SCS can show evidence to improve motor deficits in people with Type 2, 3, or 4 spinal muscular atrophy (SMA). The investigators will enroll up to six subjects with Type 2, 3, or 4 SMA aged 16 or older that show quantifiable motor deficits of the upper body. The investigators will then implant the subjects with percutaneous, linear spinal leads near the cervical spinal cord for a period of up to 29 days. Although these leads are not optimized for motor function but rather for their clinically approved indication of treating pain, the investigators believe they provide a safe technology enabling our team to perform scientific measurement necessary to evaluate potential for effects of SCS in motor paralysis with SMA. After the end of the study, the leads will be explanted.

DETAILED DESCRIPTION:
The investigators plan to 1. verify that spinal cord stimulation increases elbow muscle strength in subjects with SMA, 2. verify that spinal cord stimulation improves motor control in subjects with SMA, 3. verify that spinal cord stimulation induces measurable changes in spinal circuits and motoneuron recruitment properties in the 29 day course of implantation.

ELIGIBILITY:
SMA Participant Inclusion Criteria:

1. Subject has a diagnosis of 5q-autosomal recessive SMA confirmed by determination of a genetic deletion in the SMN1 gene (5q12.2-q13.3).
2. Subject is diagnosed as being non-ambulatory SMA based on the following criteria:

   a. Can't stand independently.
3. Subject is ≥16 years of age and < 65 years of age.
4. Subject is able to sit independently.
5. A minimum score of 1 for Entry Item "A" of the Revised Upper Limb Module (RULM) scale for SMA: "Can use hands to hold pencil or pick up a coin/token or drive a powered chair, use phone key pad"
6. Subject (and subject's parent or legal guardian if subject is a minor) is willing and able to comply with scheduled visits and study procedures
7. Participants must have started SMN inducing therapies (Spinraza or risdisplam) at least 6 months prior to enrollment. (They must have either gotten their first injection at at least 6 months prior, or they started daily intake of risdisplam at least 6 months prior to the study)

Healthy Control Participant Inclusion Criteria:

1. Subject is ≥18 years of age and < 65 years of age.
2. Subject is able to stand independently for ≥3 seconds.
3. Subject is willing and able to comply with scheduled visits and study procedures.

SMA Participant Exclusion Criteria:

1. Subject has deformation of the spinal canal preventing lead implantation as judged by the study neurosurgeon
2. Subject has size of spinal canal that is insufficient for lead implantation as judged by the study neurosurgeon
3. Subject has moderate or severe joint contractures that would affect ability to perform study measures, determined by the study physician
4. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator
5. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety of anesthesia or the procedures, make it unlikely that intervention or follow-up will be correctly completed or impair the assessment of study results, in the opinion of the investigator
6. Female subjects are pregnant or breastfeeding, as established by self-report.
7. Subject has severe claustrophobia
8. Subject is on anticoagulant, anti-spasticity or anti-seizure medication within 4 weeks of lead implantation or requires these medications during the treatment phase of the study
9. Subject has medical implant that precludes magnetic resonance imaging
10. Subject has a deconditioned respiratory system, per the discretion of the physician investigator.
11. Subjects with renal insufficiency at the discretion of the physician investigator.
12. Subjects requiring any form of sedation for MRI will be excluded.

Healthy Control Participant Exclusion Criteria:

1. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator would impact participation in the study.
2. Participants who have any serious disease or disorder (e.g. cancer, severe cardiac or respiratory disease, neurological conditions other than stroke, etc.) or cognitive impairments that could affect their ability to participate in this study.
3. Female subjects are pregnant or breastfeeding, as established by self-report.
4. Subjects requiring sedation for MRI will be excluded.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Muscle Weakness Torque | 29 days
  Isometric torque: measure the isometric torque produced by the subject at the elbow during flexion. The investigators will use the measurement of isometric torque to determine the changes in muscle strength for each participant with SCS on and with SCS off. This comparison will also include testing the non-affected arm to give the investigators a baseline for normal movement of the joint being tested. Success Criteria: ≥30% increased torque production over the SCS-off/non-affected baseline as measured during single-joint isometric torque.
Number and Severity of Adverse Events | 29 days
  Success Criteria: no serious adverse events related to the stimulation or intolerable. adverse events reported

SECONDARY OUTCOMES:
Muscle Weakness Muscle Activation | 29 days
  Muscle activation: measure surface electromyogram (EMGs) produced by the subjects during isometric movements of the elbow in the HUMAC Norm and compare to SCS-on with SCS-off and non-affected SCS side performances. Meaningful Change: >20% EMG root-mean-square (RMS) compared to SCS-on.
Motor Function ROM | 29 days
  Range of Motion (ROM): Meaningful Change: Increase of >20% of the elbow joint (if available) during SCS-on against SCS-off and SCS-non affected arm as measured by the HUMAC Norm during single-joint isotonic trials.
Motor Function RULM | 29 days
  The Revised Upper Limb Module (RULM) for SMA is a further refined version of the Hammersmith Functional Motor Scale Extended and includes specific items focused on upper-limb motor control such as raising the arms above the head that are particularly relevant for the Type 2 population of the study, or those with further progressed Type 3 and Type 4. The scale is a performance evaluation with a total score ranging from 0, if none of the activities is achieved, to 37, if all the activities are achieved fully, so a higher score means a better outcome. For our study, we require participants to score at least a 4 to be eligible. Meaningful Change: ≥2 point improvement. Compare outcomes between SCS-on and SCS-off as well as the non-affected arm.
Motor Function Fatigue | 29 days
  Fatigue will be assessed during motor function tests. Patients will be asked to provide a score from 1-10, where a greater number indicates a greater amount of fatigue for each stimulation configuration.
Discomfort/Pain | 29 days
  Patients will be asked to provide a score from 1-10, where a greater number indicates a greater amount of discomfort for each stimulation configuration. Spinal cord stimulation produces tingling sensations and other type of sensory phenomena. It is important to document that stimulation intensities required to improve motor function remain within a range of non-painful sensations.
Sensorimotor Network Structure Density | 29 days
  The investigators will perform high-definition weighted imaging to quantify fractional anisotropy as a measurement of axon density in the brain and spinal cord pre and post study.
Impression | 29 days
  The investigators will collect subjects and therapist feedback on how the technology is performing and what they would want to modify using The Clinical Global Impression Scale, a scale of 1-7 where a lower number indicates better performance and a higher number indicates more greatly impacted by their disease.
Sensorimotor Network Structure Integrity | 29 days
  The investigators will perform high-definition diffusion weighted imaging to quantify fractional anisotropy as a measurement of axon integrity in the brain and spinal cord pre and post study.
Sensorimotor Network Function | 29 days
  The investigators will perform resting state and motor-task functional MRI of the brain and spinal cord to quantify neural network activation at rest and during the execution of simple motor task such as leg muscle contraction.
Cortico-spinal Tract Integrity | 29 days
  The investigators will measure muscle evoked potential consequent to Transcranial Magnetic Stimulation of the cortico-spinal tract to assess the integrity of the cortico-spinal tract.
Spinal Circuit Excitability | 29 days
  The investigators will measure H-reflexes of the arm muscles to quantify excitability of spinal motoneurons to stimulation of primary sensory afferents pre and post-study. Expected Result: Our main scientific hypothesis is that SCS will restore monosynaptic responses of weak spinal motoneurons, thus increasing H-reflex responses pre and post study.
Motoneuron Firing Rates | 29 days
  The investigators will use high-density EMGs on leg muscles to calculate firing rates of single spinal motoneuron discharge during isometric maximal voluntary contractions.
Motor Firing Number | 29 days
  The investigators will use high-density EMGs on arm muscles to calculate the number of firing rates of single spinal motoneuron discharge during isometric maximal voluntary contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Capogrosso, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 2 years from enrollment of first participant.
Access Criteria: Data must be directly requested to the PI and will be shared upon completion of necessary data sharing agreement to protect confidential patient information.